CLINICAL TRIAL: NCT04821752
Title: Non-Persistent Environmental Toxicants Avoidance Study for Individuals With Glucose Dysregulation Who Are Not Using Insulin (NPETA-GD)
Brief Title: Environmental Toxicants Avoidance Study
Acronym: NPETA-GD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Laboratory resource constraints
Sponsor: Bastyr University (Other)
Responsible Party: Principal Investigator, Paola Costa-Mallen, Associate Research Scientist, Bastyr University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-1672
Record Dates: First submitted 2021-03-22; First posted 2021-03-30 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Pollution; Exposure; Glucose Intolerance; Glycemic Control
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: This is a single-arm trial with rolling enrollment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toxicant avoidance and glucose dysregulation (Experimental): To investigate whether or not the excretion of urinary toxicant metabolites is reduced by dietary modification and lifestyle intervention in people with glucose dysregulation; whether the participant's ranked glucose dysregulation correlates with the amount and/or type of toxic metabolites excreted at baseline; and whether the body's immediate response to glucose is improved by the reduction of toxicant burden.
  Interventions: Behavioral: Avoidance Education

INTERVENTIONS:
Behavioral: Avoidance Education — Reduction of environmental toxins exposure from the diet will be achieved by switching to organic foods. Reduction of residential and occupational exposure to toxins from household cleaning products, cosmetics, personal care products, and other sources will be achieved by switching to safer products or avoidance of the toxic exposure.

SUMMARY:
This study is designed to test whether non-persistent environmental chemicals (PECs) are elevated in people with glucose dysregulation. The primary aim is to measure whether this toxicant burden can be reduced using a dietary and lifestyle modification intervention. The secondary aim is to observe any changes in glucose response pre and post-intervention.

DETAILED DESCRIPTION:
The primary aim will be measured using a commercially-available screening test for urinary toxicant metabolites. The toxicant burden will be measured by a percentile score of each metabolite and summing all percentile values. A risk level of each metabolite will be normalized by the percentile score in order to calculate the total toxic burden for an individual. Wilcoxon-ranked sum non-parametric calculations will be used to evaluate whether pre and post-intervention reduction has occurred. Because this is a single-arm trial, any reduction in the toxicant burden will be correlated with the relative improvement of the secondary endpoint and will be measured using Kendall's tau-beta ranked correlation.

The secondary aim will assess each participant's fasting and post-prandial glucose response measured daily for throughout the 3-week trial. Because this study is not powered, the estimated man reduction from baseline cannot be estimated. Any reduction in blood glucose mean values will allow us to calculate an effect size for future investigation. The ranking of the improvement in glucose response (AUC) will be tested by ranking the reduction of the toxic burden by a correlation analysis using Kendall's tau-beta ranked correlation described above.

Each participant is provided with a baseline in-person assessment, one midpoint education session and a final assessment session. Each participant will receive a standardized packet of information regarding dietary and lifestyle interventions which reduce toxicant exposures along with a water filter for home use and gift card to support the purchase of organic food during the trial. Questionnaires including a Medical Symptom Questionnaire, Weekly Stress Inventory and Knowledge Attitudes and Behavior Questionnaire will be administered pre and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Able to complete the remote informed consent process.
3. Glucose dysregulation with HbA1c >= 5.7% at baseline
4. If hemoglobin A1c (HgA1c) is greater than 6.5% and the potential participant is not already receiving standard care for diabetes from a physician, participants must see their primary care provider for diabetes standard care before enrollment in the study.
5. Those not already eating a majority organic-food diet and drinking filtered water (>50% by self-disclosure)

Exclusion Criteria

1. Use of insulin or insulin analog medications
2. Planning to have elective surgery, diagnostic procedures, dental, or cosmetic procedures during the study period
3. Unable or unwilling to modify dietary and lifestyle behaviors
4. Those already eating a majority organic-food diet and drinking filtered water (>50% by self-disclosure)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in percentile score of urinary excretion of toxicant marker metabolites pre and post three-week dietary and lifestyle intervention | 3 months
  The primary aim will be measured using a commercially-available screening test for urinary toxicant metabolites. The toxicant burden will be measured by a percentile score of each metabolite and summing all percentile values. A risk level of each metabolite will be normalized by the percentile score in order to calculate the total toxic burden for an individual. Wilcoxon-ranked sum non-parametric calculations will be used to evaluate whether pre and post-intervention reduction has occurred. Because this is a single-arm trial, any reduction in the toxicant burden will be correlated with the relative improvement of the secondary endpoint and will be measured using Kendall's tau-beta ranked correlation.

SECONDARY OUTCOMES:
Change in immediate glucose response measured by daily fasting and post-prandial blood glucose measurements. | 3 months
  A secondary endpoint is to observe each participant's glucose response throughout the 3-week trial period. Because this is not powered, the estimated mean reduction from the baseline to the ending of the trial cannot be estimated. Any reduction in the blood glucose mean values allows us to calculate the effect size for future investigation. The ranking of the improvement in glucose response (smaller AUC) is tested with the ranking of the reduction of toxic burden by a correlation analysis described the above.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Costa-Mallen, PhD, Principal Investigator — Bastyr University
Locations (1):
- Bastyr University, Kenmore, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in any publications, after deidentification (text, tables, figures and appendices).
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).